CLINICAL TRIAL: NCT05475574
Title: Impact of Discontinuing Contact Precautions for Extended-spectrum β-lactamase Enterobacteriaceae (ESBLE) in a Geriatric Unit: an Interventional Prospective Noninferiority Non-randomized Double-blind Controlled Before and After Study
Brief Title: Impact of Discontinuing Contact Precautions for Extended-spectrum β-lactamase Enterobacteriaceae in a Geriatric Unit
Acronym: Ger-SP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 2021-05-CHRMT
Record Dates: First submitted 2022-07-13; First posted 2022-07-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Infection, Hospital
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Before discontinuation of contact precautions for ESBLE (No Intervention): Implementation of contact precaution in addition to standard precaution for any patient carrying (infected or colonized) ESBLE
- After discontinuation of contact precautions for ESBLE (Experimental): Discontinuation of contact precaution : only standard precaution are implemented for any patient carrying (infected or colonized) ESBLE
  Interventions: Other: Discontinuation of contact precautions for ESBLE

INTERVENTIONS:
Other: Discontinuation of contact precautions for ESBLE — Discontinuation of contact precaution : only standard precaution are implemented for any patient carrying (infected or colonized) ESBLE
  Arms: After discontinuation of contact precautions for ESBLE

SUMMARY:
This is an interventional multicenter prospective noninferiority non-randomized double-blind controlled before and after study.

The aim of this study is to demonstrate that standard precautions alone are not inferior to contact precautions by comparing the incidence density of extended-spectrum β-lactamase (ESBL)-producing Enterobacteriaceae acquired in geriatric units before and after discontinuing contact precautions.

DETAILED DESCRIPTION:
Healthcare-associated infections (HAIs) are one of the main causes of morbidity and mortality worldwide. Extended-spectrum β-lactamase (ESBL)-producing Enterobacteriaceae have become microorganisms frequently found in HAIs, which reduces the therapeutic possibilities.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (> 65 years old)
* Patient hospitalized in geriatrics during the study period
* Free and informed consent obtained from the patient (or his trusted person or legal representative) within 48 hours of its admission at the geriatric unit
* Patient affiliated to a social security scheme

Non Inclusion Criteria:

* Patient requiring contact precaution for an indication other than ESBLE (COVID-19, classical PCC excluding EBLSE, Clostridium difficile PCC, scabies PCC and BHRe PCC) on admission
* Patient under legal protection
* Person deprived of liberty

Exclusion criteria:

* Patient requiring contact precaution for an indication other than ESBL during the patient stay (COVID-19, classical PCC excluding EBLSE, Clostridium difficile PCC, scabies PCC and BHRe PCC)
* Patient's stay period less than 4 days

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 954 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2029-09-07 (Estimated); Study Completion 2029-09-21 (Estimated)

PRIMARY OUTCOMES:
Incidence density of acquired ESBLE | during 6 month period
  Incidence density of acquired ESBLE in geriatric unit for 1000 days of hospitalization is calculated by dividing the number of acquired ESBLE by the number of days of patients' hospitalization multiplied by 1000 Acquisition of ESBLE is defined by a positive sample in patient on discharge day with a negative sample on admission in geriatric unit A positive sample is defined by the presence of at least one ESBLE on a clinical (infection) or screening (colonization) sample.
  The hospitalisation number is calculated as the cumulative length of stay of all patients at risk (= negative on admission).

SECONDARY OUTCOMES:
Incidence density of acquired ESBLE by species during 6 month period | during 6 month period
  Incidence density of acquired ESBLE in geriatric unit by species (E. coli versus non-E. coli) for 1000 days of hospitalization. This is calculated by dividing the number of acquired ESBLE by species by the number of days of patients' hospitalization multiplied by 1000.
  Acquisition of ESBLE is defined by a positive sample in patient on discharge day with a negative sample on admission in geriatric unit A positive sample is defined by the presence of at least one ESBLE on a clinical (infection) or screening (colonization) sample.
  The hospitalisation number is calculated as the cumulative length of stay of all patients at risk (= negative on admission).
The rate of compliance with hand hygiene in health care providers | Up to 3 months per health department
  The evaluation of the compliance with hygiene measures is calculated in health care providers by dividing the number of hand hygiene moments carried out by the number of opportunities multiplied by 100, according to the World Health Organization (WHO) methodology
Evaluation of the barriers to alcohol-based hand rub in case of non-compliance in health care providers | Up to 3 months per health department
  The barriers to alcohol-based hand rub are identified in case of non-compliance, using a Pulpe' friction questionnaire (RéPIAS) where professionals are interviewed about their practices in terms of hand hygiene. For each situation, the professional is also asked how important it is for him to perform hand hygiene in each situation listed above, with a slider to be positioned between 0 (not at all important; worse outcome) and 10 (the most important; better outcome).
The rate of compliance with personal protective equipment | Up to 3 months per health department
  The rate of compliance with the wearing and removal of personal protective equipment throughout patient care, is observed during care related to the management of excreta (changing, putting on or removing a dish basin, use of a basin washer-disinfector).
  The rate is calculated by dividing the number of personal protective equipment good caring practices by the number of opportunities multiplied by 100.
Evaluation of satisfaction related to patient care, by self-questionnaire Hospital anxiety and depression scale (HADS) | on the day of discharge of the geriatric unit, on average on the 11th day
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item measure designed to assess anxiety and depression symptoms in medical patients, with emphasis on reducing the impact of physical illness on the total score.
  Items are rated on a 4-point severity scale. The HADS produces two scales, one for anxiety (HADS-A) and one for depression (HADS-D), differentiating the two states. Scores of greater than or equal to 11 on either scale indicate a definitive case.

CONTACTS AND LOCATIONS:
Overall Officials: Noel BLETTNER, MD, Principal Investigator — Mercy Hospital CHR Metz Thionville; Azzeddine AZZEMOU, MD, Principal Investigator — Bel Air Hospital CHR Metz Thionville
Locations (1):
- CHR Metz-Thionville/Hôpital Bel Air, Metz, France